CLINICAL TRIAL: NCT05605964
Title: Relugolix Versus Leuprolide in Patients With Prostate Cancer: A Randomized, Open-Label Study to Assess Major Adverse Cardiovascular Events (REPLACE-CV)
Brief Title: Randomized Study to Evaluate MACE in Patients With Prostate Cancer Treated With Relugolix or Leuprolide Acetate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MVT-601-056
Record Dates: First submitted 2022-10-25; First posted 2022-11-04 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: ORGOVYX; relugolix; prostate cancer; leuprolide acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — relugolix; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Relugolix (Experimental): Oral relugolix 120 mg once daily with a loading dose of 360 mg on Day 1
  Interventions: Drug: Relugolix
- Leuprolide Acetate (Active Comparator): Subcutaneous or intramuscular leuprolide acetate 22.5 mg 3-M depot or 45 mg 6-M injection or Leuprolide acetate injectable emulsion (42 mg injectable emulsion is not allowed)
  Interventions: Drug: Leuprolide Acetate

INTERVENTIONS:
Drug: Relugolix — Relugolix tablet
  Other Names: ORGOVYX; TAK-385; MVT-601; RVT-601; T-1331285
  Arms: Relugolix
Drug: Leuprolide Acetate — Leuprolide acetate injection
  Other Names: Leuprolide
  Arms: Leuprolide Acetate

SUMMARY:
This was a randomized study to evaluate the risk of major adverse cardiovascular events (MACE) for relugolix compared with leuprolide acetate. Enrollment in this study was discontinued by the Sponsor on 01 Dec 2023. In an effort to mitigate any treatment interruptions, actively enrolled patients will be allowed to remain on study drug up to a period of 12 months ending Dec 2024 if they choose to remain in the discontinuation phase of the study.

DETAILED DESCRIPTION:
Eligible patients were randomized (1:1) to receive either relugolix or leuprolide acetate for prostate cancer or as an adjunct to primary or salvage radiation therapy. The study was intended to collect clinical and cardiovascular risk factor data on patients ages 18 and older who were receiving relugolix or leuprolide acetate for their prostate cancer or as adjunct to radiation therapy with a treatment plan to be on at least 12 months of continuous ADT. Enrollment in this study was discontinued by the Sponsor on 04 Dec 2023. In an effort to mitigate any treatment interruptions, actively enrolled patients will be allowed to remain on study drug up to a period of 12 months ending Dec 2024. During this discontinuation phase, all active investigative sites will be expected to formulate a transition plan for their study patients from this clinical study to SOC as soon as practicable.

The primary endpoint in this study was the time to first adjudicated MACE (nonfatal myocardial infarction, nonfatal stroke, and cardiovascular death). However, with the discontinuation of enrollment in the study on 04 DEC 2023 by the sponsor, the primary endpoint will be to describe the safety of relugolix in the study population while actively enrolled patients remain on study drug.

ELIGIBILITY:
A patient will be eligible for inclusion in the discontinuation phase of the study if the following applies:

1. Was previously enrolled under the original version and amendment 1 of this study
2. Has voluntarily resigned and dated the informed consent form prior to transition to the discontinuation phase of this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Safety Outcomes | Screening; Day 1; 3, 6, 9, and 12 months; and every 3 months thereafter
  Incidence of selective safety data including all serious adverse events, nonserious adverse events leading to discontinuation of relugolix or leuprolide acetate, and clinical laboratory tests as obtained per standard of care

CONTACTS AND LOCATIONS:
Locations (104):
- United States (104):
  - Urology Associates of Mobile, Mobile, Alabama
  - Arizona Urology Specialists, PLLC, Tucson, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Genesis Research, LLC Satellite, Downey, California
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - Genesis Research , LLC, Los Alamitos, California
  - Tower Urology, Los Angeles, California
  - Pacific Cancer Care, Monterey, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Tri Valley Urology Medical Group Satellite, Murrieta, California
  - San Bernadino Urological Associates Medical Group, San Bernardino, California
  - Genesis Research, LLC, San Diego, California
  - Genesis Research, LLC Satellite, Sherman Oaks, California
  - Tri Valley Urology Medical Group Satellite, Temecula, California
  - Genesis Research, LLC Satellite, Torrance, California
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Urologic Surgeons of Washington, Washington D.C., District of Columbia
  - Advanced Urology Institute, Daytona Beach, Florida
  - East Coast Institute for Research, LLC Satellite, Jacksonville, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Lake City Cancer Center, LLC, Lake City, Florida
  - SG Research LLC, Miami, Florida
  - Florida Urology Partners, LLP Satellite, Tampa, Florida
  - Florida Urology Partners, LLP, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Georgia Cancer Center Satellite, Augusta, Georgia
  - St. Luke's Regional Medical Center Satellite, Boise, Idaho
  - St. Luke's Regional Medical Center, Boise, Idaho
  - St. Luke's Cancer Institute - Fruitland Satellite, Fruitland, Idaho
  - St. Luke's Cancer Institute - Meridian Satellite, Meridian, Idaho
  - St. Luke's Meridian Medical Center Satellite, Meridian, Idaho
  - St. Luke's Cancer Institute - Nampa Satellite, Nampa, Idaho
  - St. Luke's Nampa Medical Center Satellite, Nampa, Idaho
  - St. Luke's Cancer Institute Satellite, Twin Falls, Idaho
  - St. Luke's Magic Valley Medical Center Satellite, Twin Falls, Idaho
  - Illinois CancerCare - Bloomington Satellite, Bloomington, Illinois
  - Northwestern University, Chicago, Illinois
  - Swedish Hospital Satellite, Chicago, Illinois
  - Associated Urological Specialists, Chicago Ridge, Illinois
  - NorthShore University Health System - Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare - Galesburg Satellite, Galesburg, Illinois
  - NorthShore University Health System - Glenbrook Hospital Ambulatory Care Center Satellite, Glenview, Illinois
  - NorthShore University Health System - Highland Park Hospital Ambulatory Care Center Satellite, Highland Park, Illinois
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - Advanced Urology Associates, New Lenox, Illinois
  - Illinois CancerCare - Ottawa Satellite, Ottawa, Illinois
  - Illinois CancerCare - Pekin Satellite, Pekin, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Illinois CancerCare - Peru Satellite, Peru, Illinois
  - Illinois CancerCare - Washington Satellite, Washington, Illinois
  - Urology of Indiana, LLC Satellite, Carmel, Indiana
  - Urology of Indiana, LLC, Greenwood, Indiana
  - IU Health Arnett Cancer Center, Lafayette, Indiana
  - IU Health Ball Memorial Hospital Satellite, Muncie, Indiana
  - Adult and Pediatric Urology P.C. Satellite, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Wichita Urology Group Satellite, Wichita, Kansas
  - Wichita Urology Group, Wichita, Kansas
  - Comprehensive Urology, Royal Oak, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - Lake Regional Health System, Osage Beach, Missouri
  - Specialty Clinical Research of St. Louis, St Louis, Missouri
  - Urology of St. Louis Satellite, St Louis, Missouri
  - St. Vincent Healthcare Satellite, Billings, Montana
  - St. Vincent - Frontier Cancer Center, Billings, Montana
  - Adult and Pediatric Urology P.C., Omaha, Nebraska
  - Capital Health Medical Center - Hopewell, Pennington, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Associated Medical Professionals of NY, PLLC, Syracuse, New York
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Altru Cancer Center, Grand Forks, North Dakota
  - Altru Health System Satellite, Grand Forks, North Dakota
  - Altru Professional Center Satellite, Grand Forks, North Dakota
  - University Hospitals Seidman Cancer Center at UH Avon Health Center Satellite, Avon, Ohio
  - TriState Urologic Services PSC Inc., Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Central Ohio Urology Group Satellite, Gahanna, Ohio
  - Central Ohio Urology Group, Gahanna, Ohio
  - University Hospitals Seidman Cancer Center at UH Mentor Health Center Satellite, Mentor, Ohio
  - Helios CR, LLC, Middleburg Heights, Ohio
  - UH Minoff Health Center at Chagrin Highlands, Orange, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - Robert Packer Hospital Satellite, Sayre, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Lowcountry Urology Clinics, North Charleston, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Valley Cancer Associates, Harlingen, Texas
  - Houston Metro Urology CRC, LLC, Houston, Texas
  - Urology San Antonio Clinical Trials, San Antonio, Texas
  - The Urology Place, San Antonio, Texas
  - Logan Regional Hospital Satellite, Logan, Utah
  - Intermountain Medical Center Satellite, Murray, Utah
  - McKay-Dee Hospital Satellite, Ogden, Utah
  - Utah Valley Hospital, Provo, Utah
  - St. George Regional Hospital Satellite, St. George, Utah
  - Potomac Urology Center, PC, Alexandria, Virginia
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - Potomac Urology Satellite, Woodbridge, Virginia
  - Spokane Urology, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No